CLINICAL TRIAL: NCT00150085
Title: A Prospective, Randomized, Open-label, Twenty-six Week Study of the Efficacy and Safety of Converting Kidney and Liver Transplant Recipients With Tacrolimus-associated Abnormal Glucose Metabolism to Cyclosporine Micro-emulsion With C2 Monitoring
Brief Title: Safety and Efficacy of Converting Maintenance Kidney and Liver Transplant Recipients With Abnormal Glucose Metabolism From Tacrolimus to Cyclosporine Micro-emulsion
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Novartis, Novartis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COLO400AUS06
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2011-02

CONDITIONS: Tacrolimus-associated Abnormal Glucose Metabolism in Kidney and Liver Transplant Recipients
Keywords: diabetes, glucose, tacrolimus, cyclosporine micro-emulsion, liver, kidney, renal
MeSH Terms: conditions — Diabetes Mellitus

INTERVENTIONS:
Drug: cyclosporine micro-emulsion

SUMMARY:
New onset diabetes mellitus (NODM) post- transplantation decreases patient and graft survival. Some immunosuppressive agents are associated with a higher incidence of NODM. This study evaluates the safety and efficacy of converting patients with NODM from tacrolimus to cyclosporine micro-emulsion as a primary immunosuppressant for kidney and liver recipients.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of first or second cadaveric or living donor kidney transplantation or first cadaveric or living donor liver transplantation
* Receiving tacrolimus as a primary immunosuppressant
* Currently on any diabetic agent or meets the American Diabetes Association definition of diabetes mellitus

Exclusion Criteria:

* History of treated diabetes mellitus prior to transplantation
* Less than 2 weeks post-transplantation for kidney and less than 8 weeks for liver
* Greater than 36 months post-transplantation
* Onset of diabetes is greater than 12 months prior to time of study entry
* Has unacceptable or unstable graft function

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-02; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who no longer require a hypoglycemic agent, or who move from insulin to an oral agent, or who no longer meet the American Diabetes Association criteria, or a relative improvement in mean glycosylated hemoglobin at 12 and 26 weeks

SECONDARY OUTCOMES:
Safety assessed by death, graft loss, biopsy supported clinically manifested acute rejection, change in kidney function, change in liver function, serious adverse events and adverse events at 12 and 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis